CLINICAL TRIAL: NCT06456853
Title: Comparison of AI-Generated Pain Scoring Visuals With Visual Analog Scale (VAS) for Pain Assessment
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Engin Ihsan Turan, anesthesiology and reanimation specialist, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: AI Images
Record Dates: First submitted 2024-06-08; First posted 2024-06-13 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Pain, Postoperative
Keywords: Postoperative Pain; Artificial Intelligence; Pain assesment
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Visual Analog Scale Score: The Visual Analog Scale (VAS) pain score is a simple and effective method used to measure patients' pain levels. This method is typically represented by a line ranging from 0 to 10, where 0 indicates no pain and 10 indicates the most severe pain. Patients are asked to mark a point on the line that corresponds to their level of pain.
  Interventions: Other: Pain assesment
- Images maded by Artificial Intelligence: Pain assesment maded by images which is created from ChatGPT/DALLE
  Interventions: Other: Pain assesment

INTERVENTIONS:
Other: Pain assesment — We will ask patients about their pain and will try to asses their pain scores. Then we will ask them to which methot is more suitable for assesment.

SUMMARY:
This prospective study will be conducted in surgical wards, assessing postoperative patients. Initially, patients will be evaluated using the VAS method. Subsequently, they will be shown five AI-generated images depicting different pain levels and will select the image that best represents their pain. A follow-up survey will assess the effectiveness of each method.

Using ChatGPT-4/DALL-E, images corresponding to VAS scores of 1-2, 3-4, 5-6, 7-8, and 9-10 will be created. Patients will choose the image that best describes their pain, aiming to determine if AI-supported visuals offer a more accurate alternative to VAS for pain assessment.

DETAILED DESCRIPTION:
Study Objective The primary objective of this study is to compare and evaluate the effectiveness of AI-generated pain visuals in assisting patients to express their pain levels with the Visual Analog Scale (VAS). By allowing patients to more accurately depict their pain through AI-supported visuals, the study aims to enhance pain management practices in clinical settings.

Study Significance Pain management is a critical component of healthcare, directly impacting patient well-being and treatment success. The VAS is a widely used tool for subjective pain assessment but can be challenging for some patients due to its abstract nature. AI-generated visuals offer a potentially more precise and understandable way for patients to communicate their pain, potentially leading to more accurate and personalized pain assessments and management.

This study aims to measure the contribution of AI-generated pain visuals to more accurate pain assessment and to explore the potential applications of this technology. Additionally, the study seeks to understand the advantages and limitations of this approach compared to traditional methods like VAS, thereby enhancing the role of AI in pain management practices.

Expected Benefits and Risks

Expected Benefits:

Improved Pain Expression: AI-generated visuals may help patients articulate their pain more clearly, leading to better pain management in clinical settings.

Personalized Treatment Approaches: Enhanced pain expression can provide healthcare providers with opportunities to create more personalized treatment plans, especially beneficial for chronic pain patients.

Enhanced Clinical Decision-Making: The use of AI visuals may facilitate more objective and reproducible pain assessments, improving overall pain management strategies.

Potential Risks:

Misinterpretation Risk: AI-generated visuals might misinterpret patient pain in certain cases, especially if the visuals are misleading or complex.

Dependence on Technology: Over-reliance on AI tools may overlook the importance of human judgment and the subjective nature of pain assessment.

Study Design This prospective study will be conducted in surgical wards, assessing postoperative patients. Initially, patients will be evaluated using the conventional VAS method, which involves marking their pain on a 0-10 scale. Subsequently, patients will be shown five AI-generated images depicting different pain levels and asked to select the image that best represents their pain. A follow-up survey will assess which method the patients found more effective for expressing their pain.

VAS Scoring:

Patients will mark their pain level on a line ranging from 0 (no pain) to 10 (worst pain).

AI-Generated Visuals:

Using ChatGPT-4/DALL-E, images corresponding to VAS scores of 1-2, 3-4, 5-6, 7-8, and 9-10 will be created. These images will specifically depict facial expressions reflecting the respective pain levels. Patients will choose the image that best describes their pain.

This study aims to identify whether AI-supported visuals provide a more accurate and user-friendly alternative to traditional VAS scoring for pain assessment.

VAS Score Descriptions VAS Score 1-2: A middle-aged man showing signs of mild discomfort.

VAS Score 3-4: A young female athlete on a soccer field expressing moderate pain.

VAS Score 5-6: A man in a kitchen environment displaying severe pain from a cut.

VAS Score 7-8: A young male feeling severe shoulder pain.

VAS Score 9-10: A young woman experiencing intense pain.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above
* Underwent surgery for any reason
* Consented to participate in the study and signed the informed consent form

Exclusion Criteria:

* Patients under 18 years old
* Patients who did not sign the informed consent form
* Patients with visual impairments
* Patients whose level of consciousness is not sufficient to complete the survey
* Patients with a history of psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: VAS scoring and pain assessment using visuals will be conducted on at least 398 patients aged 18 and above who have undergone any surgery, at any time within the first 24 hours postoperatively.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2024-06-14 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
Pain assesment | 10 minutes
  The primary outcome for this research is to compare the effectiveness of AI-generated pain assessment visuals with the traditional Visual Analog Scale (VAS) in accurately evaluating and expressing patients' pain levels. This will be measured through patient-reported ease of use, clarity, and usefulness of both methods, as well as patient preference for either method in pain assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All patients IPD will delete and we will give randomised patient number to them